CLINICAL TRIAL: NCT00936338
Title: Randomized Clinical Trial of Treatment for Temporomandibular Joint (TMJ) Disc Displacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Herniated Disk; Temporomandibular Disorders
Keywords: anterior disc displacement without reduction of temporomandibular disorders
MeSH Terms: conditions — Intervertebral Disc Displacement; Temporomandibular Joint Disorders | interventions — Splints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- splint (Active Comparator)
  Interventions: Behavioral: splint and joint mobilization self exercise
- joint mobilization self exercise (Active Comparator)
  Interventions: Behavioral: splint and joint mobilization self exercise

INTERVENTIONS:
Behavioral: splint and joint mobilization self exercise

SUMMARY:
The effectiveness of physical therapy for treatment of anterior disc displacement without reduction of temporomandibular disorders has not been well defined. This study compared the treatment method with conservative splint therapy. Fifty two subjects were assigned at random to either of two treatment groups: one is a splint treatment group, and the other is a joint mobilization self exercise group. Each treatment was evaluated using four outcome variables: (i) maximum mouth opening range without and (ii) with pain, (iii) present pain intensity, and (iv) limitation of daily activities. All outcome variables were significantly improved after eight-week of treatment in the exercise group. Meanwhile, the splint treatment improved three variables, other than "mouth opening with pain"; however, the degree of improvement was less than that seen in the exercise group. This result demonstrates that the joint mobilization self exercise improves jaw function and relieves pain as compared to the splint treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) male or female over 18 years old;
* (2) with mouth opening pain on the TMJ affected side;
* (3) over two weeks after the onset of ADDwoR;
* (4) with maximum mouth opening of less than 40 mm; and
* (5) MRI-confirmed ADDwoR. The

Exclusion Criteria:

* (1) unwilling or unable to receive splint and/or exercise therapy;
* (2) with systemic bone or joint disease,
* (3) regular medication such as analgesics, anti-anxiety drugs, antidepressants and psychotropics; and
* (4) missing teeth and/or a removable denture but having a fixed partial denture restoration over one year.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
(i) maximum mouth opening range without and (ii) with pain, (iii) present pain intensity, and (iv) limitation of daily activities | 0, 4 and 8 week

CONTACTS AND LOCATIONS:
Locations (1):
- TMJ Clinic, Tokyo Medical and Dental University, Tokyo, Japan